CLINICAL TRIAL: NCT06962488
Title: Clinical Implementation of Blood Pressure Polygenic Risk Score
Brief Title: Polygenic Risk Score Implementation and Stratification for Managing Blood Pressure
Acronym: PRISM-BP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Pankaj Arora, MD, Associate Professor, Division of Cardiovasular Disease, Department of Medicine, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB-300014760; R01HL176882 (NIH)
Record Dates: First submitted 2025-04-21; First posted 2025-05-08 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Hypertension; Atherosclerotic Cardiovascular Disease
Keywords: Systolic Blood Pressure; Polygenic Risk Score; Genomic Counseling; Health Belief Model; Cardiovascular Health
MeSH Terms: conditions — Hypertension; Atherosclerosis; Genetic Risk Score

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SBP PRS Dissemination (Experimental): Participants randomized to this arm will receive their personalized SBP polygenic risk score (PRS), along with structured genomic counseling sessions guided by the Health Belief Model and routine clinical care. Counseling will be delivered by trained genetic counselors at baseline and during 3-monthly in-person follow-up visits. The counseling is designed to increase perceived susceptibility, reduce perceived barriers, and improve self-efficacy for health behavior change.
  Interventions: Behavioral: SBP PRS Dissemination
- Routine Clinical Care (Active Comparator): Participants randomized to this arm will receive standard clinical care for hypertension, including educational materials on blood pressure control, lifestyle modification, and cardiovascular health. These materials will be adapted from the American Heart Association Life's Essential 8 and the ACC preventive cardiology toolkit. Participants will not receive SBP PRS results or genomic counseling during the study. At the end-of-study visit (12 months), participants in this group will be offered their SBP PRS results and optional genomic counseling.
  Interventions: Behavioral: Regular Care

INTERVENTIONS:
Behavioral: Regular Care — Educational brochures and lifestyle guidance on blood pressure control, medication adherence, physical activity, and healthy diet, provided at baseline only. No additional counseling or genetic risk disclosure will occur during the 12-month intervention period.
  Arms: Routine Clinical Care
Behavioral: SBP PRS Dissemination — Participants receive individualized SBP PRS reports and structured genomic counseling sessions delivered by trained genetic counselors. Counseling addresses key constructs of the Health Belief Model, including perceived susceptibility, severity, and benefits of behavior change, with an emphasis on lifestyle modification and medication adherence.
  Arms: SBP PRS Dissemination

SUMMARY:
In a multi-ethnic population, a genome-wide polygenic risk score (PRS) for systolic blood pressure (SBP), incorporating over one million common genetic variants, predicts blood pressure (BP) traits and the risk of adverse cardiovascular events beyond traditional risk factors. Delivering SBP PRS information to young and middle-aged adults with hypertension (HTN) and poor cardiovascular health (CVH) may enhance their motivation to adopt healthier lifestyles, improve blood pressure control, and ultimately reduce the risk of future cardiovascular disease (CVD). This randomized controlled trial will assess the impact of SBP PRS disclosure and theory-based genomic counseling on systolic blood pressure and health behaviors. A total of 300 adults aged 18-55 years will be enrolled and randomized to receive either routine clinical care or SBP PRS results with structured genomic counseling based on the Health Belief Model (HBM). Participants will be followed for 12 months. The primary outcome is change in 24-hour mean SBP from baseline to one year. Secondary outcomes include changes in physical activity, diet, medication adherence, smoking, lipid and glucose levels, and body composition. The study will also evaluate how behavior change is influenced by health beliefs, including perceived risk and self-efficacy. This study aims to advance the use of genomic tools in hypertension management and cardiovascular disease prevention.

DETAILED DESCRIPTION:
This parallel-arm, randomized clinical trial is designed to assess the change in SBP following BP PRS dissemination and genomic counseling. Investigators will enroll 300 young and middle-aged adults (age: 18-55 years; 50% females; 50% non-White) with HTN [stratified by race, sex, and SBP PRS group (high vs. low/intermediate)] and poor CVH [American Heart Association's (AHA) Life Essential 8 Score: 0-50]. Participants will be randomized to A) routine clinical care (N=150), or B) SBP PRS dissemination (regular care + SBP PRS delivery and genetic counseling; N=150). After obtaining informed consent, the eligible participants will undergo genotyping and computation of their genome-wide SBP PRS. The SBP PRS results will be available within 10-15 days of screening. Participants will then be randomized in a 1:1 manner [stratified by sex, racial/ethnic group (White vs. non-White), and SBP PRS (high vs. low/intermediate)] to either the SBP PRS dissemination arm or the routine care arm. Participants will undergo a comprehensive baseline health assessment, including measurement of key HBM constructs, using the recently developed Attitudes and Beliefs about the CVD (ABCD) Risk Questionnaire, a 26-item instrument validated in the clinical setting with four subscales: perceived risk of heart attack/stroke, perceived benefits and intentions to exercise, healthy eating intentions, and perceived benefits and intentions to reducing smoking. Investigators will also assess the perceived severity of CVD, perceived barriers to prevention behaviors, and self-efficacy to perform preventive behaviors using subscales previously assessed for content and face validity by an expert review panel and patient focus groups. Physical activity status and sleep duration (using 7-day Actigraphy), detailed dietary history [using the United States Department of Agriculture (USDA) Healthy Eating Index and collected through the validated Nutrition Coordinating Center Nutrition Data System for Research (NCC NDSR) dietary assessment tool], health-related quality of life [using 36-Item Short Form Survey (SF-36), and the Centers for Disease Control and Prevention (CDC) Health-Related Quality of Life-14 (HRQOL-14)], medication adherence using the Medication Adherence Rating Scale (MARS), 24-hour ambulatory blood pressure monitoring (ABPM), current health behaviors (smoking, alcohol, recreational drugs), and other cardiometabolic health parameters [lipid profile, hemoglobin A1c (HbA1c), body mass index (BMI), and body composition), and anxiety [using the Beck Anxiety Inventory (BAI)].

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 55 years (inclusive) at the time of screening.
* Diagnosis of hypertension defined by 2017 ACC/AHA guidelines, as evidenced by Resting office systolic blood pressure (SBP) of 130-160 mm Hg or Resting office diastolic blood pressure (DBP) of 80-100 mm Hg or Current use of antihypertensive medication.
* Poor cardiovascular health, defined as Life's Essential 8 score <50.
* Willing and able to undergo 24-hour ambulatory blood pressure monitoring (ABPM) to confirm hypertension.
* Able to provide informed consent.

Exclusion Criteria:

* History of cardiovascular disease, including Myocardial infarction, Angina, Cardiac arrhythmia, Coronary heart disease, Heart failure, Stroke, or transient ischemic attack.
* Body mass index (BMI) <18.5 kg/m² or >45 kg/m².
* Baseline office SBP >160 mm Hg or DBP >100 mm Hg.
* Use of more than two antihypertensive medication classes.
* Not hypertensive based on 24-hour ABPM (per 2017 ACC/AHA criteria).
* Pregnant or breastfeeding.
* Estimated glomerular filtration rate (eGFR) <60 mL/min/1.73 m² (using CKD-EPI equation).
* Urine albumin-to-creatinine ratio ≥30 mg/g.
* Hepatic transaminase levels >3× the upper limit of normal.
* Significant psychiatric illness (assessed via Global Health Questionnaire-12).
* Moderate or severe anxiety (Beck Anxiety Inventory [BAI] score >16).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2030-03-31 (Estimated); Study Completion 2030-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in Mean 24-Hour Systolic Blood Pressure | 1 year
  The difference in the 24-hour mean systolic BP between the two study groups at 1 year, adjusted for baseline.

SECONDARY OUTCOMES:
Change in Physical Activity Levels | 1 year
  Physical activity levels in MET·hr-1·wk-1 estimated using 7-day actigraphy. The difference in the physical activity levels (MET·hr-1·wk-1) between the two study groups at 1 year, adjusted for baseline.
Change in Healthy Diet Index Score | 1 year
  The USDA Healthy Eating Index (HEI-2015) will be used to estimate changes in diet quality. The HEI score ranges from 0 to 100, with higher scores indicating better adherence to the Dietary Guidelines for Americans (i.e., better diet quality). The outcome measure will be the difference in HEI scores between the two study groups at 1 year, adjusted for baseline
Change in Medication Adherence | 1 year
  Medication adherence will be assessed using the Medication Adherence Report Scale (MARS-5). The MARS-5 scale has a score range from 5 to 25, with higher scores indicating better adherence. The outcome measure will be the difference in MARS-5 scores between the two study groups at 1 year, adjusted for baseline
Change in Ambulatory Blood Pressure Parameters | 1 year
  The difference in the 24-hour mean diastolic BP, daytime systolic BP, daytime diastolic BP, nighttime systolic BP, and nighttime diastolic BP between the two study groups at 1 year, adjusted for baseline.
Change in Lipid Profile | 1 year
  The difference in the low-density lipoprotein cholesterol, high-density lipoprotein cholesterol, triglyceride, and total cholesterol levels between the two study groups at 1 year, adjusted for baseline.
Change in Sleep Duration | 1 year
  The difference in the sleep duration estimated using 7-day actigraphy, between the two study groups at 1 year, adjusted for baseline.
Change in Body Mass Index | 1 year
  The difference in the body mass index between the two study groups at 1 year, adjusted for baseline.
Change in Fat Mass | 1 year
  The difference in the fat mass between the two study groups at 1 year, adjusted for baseline.
Change in Lean Mass | 1 year
  The difference in the lean mass between the two study groups at 1 year, adjusted for baseline.
Change in Health Belief Model Constructs | 1 year
  The difference in the Health Belief Model constructs, measured using standardized questionnaires, between the two study groups at 1 year, adjusted for baseline.
Change in Smoking Behavior | 1 year
  Estimated as the number of cigarettes per week. The difference in the number of cigarettes per week between the two study groups at 1 year, adjusted for baseline.
Change in Health-Related Quality of Life (SF-36) | 1 year
  Assessed using the 36-Item Short Form Survey (SF-36). The SF-36 produces scores ranging from 0 to 100, with higher scores indicating better quality of life. The difference between study groups at 1 year will be assessed, adjusted for baseline.
Change in Health-Related Quality of Life (CDC HRQOL-14) | 1 year
  Assessed using the Centers for Disease Control and Prevention Health-Related Quality of Life 14-item measure (CDC HRQOL-14). The number of physically and mentally unhealthy days is recorded, with higher numbers indicating worse quality of life. The difference between study groups at 1 year will be assessed, adjusted for baseline.
Change in Anxiety | 1 year
  Anxiety will be assessed using the Beck Anxiety Inventory (BAI). The BAI scores range from 0 to 63, with higher scores indicating greater severity of anxiety symptoms. The outcome measure will be the difference in BAI scores between the two study groups at 1 year, adjusted for baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Pankaj Arora, MD, FAHA, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shetty NS, Pampana A, Patel N, Yerabolu K, Patel G, Irvin MR, Natarajan P, Lin HJ, Guo X, Rich SS, Rotter JI, Li P, Arora G, Arora P. Sex Differences in the Association of Multiethnic Genome-Wide Blood Pressure Polygenic Risk Score With Population-Level Systolic Blood Pressure Trajectories. Circ Genom Precis Med. 2024 Apr;17(2):e004515. doi: 10.1161/CIRCGEN.123.004515. Epub 2024 Feb 19. No abstract available. PMID 38372177
- [Background] Shetty NS, Pampana A, Patel N, Li P, Yerabolu K, Gaonkar M, Arora G, Arora P. Sex Differences in the Association of Genome-Wide Systolic Blood Pressure Polygenic Risk Score With Hypertension. Circ Genom Precis Med. 2023 Dec;16(6):e004259. doi: 10.1161/CIRCGEN.123.004259. Epub 2023 Oct 9. No abstract available. PMID 37807951